CLINICAL TRIAL: NCT04223128
Title: Comparing Intravenous Single Low Doses of Magnesium Sulphate Versus Dexamethasone as Adjuvants to Ultrasound Guided Transversus Abdominis Plane (TAP) Block for Prolongation of Postcesaren Analgesia
Brief Title: Comparing Intravenous Magnesium Sulfate With Dexamethasone as Adjuvants to Ultrasound Guided TAPblock
Acronym: TAPblock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tamer Nabil Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Tamer Nabil Abdelrahman, Lecturer of anesthesia, intensive care and pain management, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: FAMSU R 59/2019
Record Dates: First submitted 2020-01-04; First posted 2020-01-10 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Group M and group D are parallel and compared to group C
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Magnesium sulfate group(M) (Active Comparator): Participants in group (M) will receive 50 mg/kg MgSO4 in 100 ml isotonic saline intravenous (I.V) over 20 minutes prior to induction of general anesthesia by 30 minutes then ultrasound guided TAPblock after closure of the abdomen
  Interventions: Procedure: Ultrasound guided transversus abdominis plane block
- Dexamethasone group(D) (Active Comparator): participants in group (D) will receive 2 mg Dexamethasone in 100 ml isotonic saline IV then ultrasound guided TAPblock after closure of the abdomen
  Interventions: Procedure: Ultrasound guided transversus abdominis plane block
- Placebo group(C) (Placebo Comparator): participants in group (C) will receive 100 ml isotonic saline IV (placebo) by the same route and over the same duration as control then ultrasound guided TAPblock after closure of the abdomen
  Interventions: Procedure: Ultrasound guided transversus abdominis plane block

INTERVENTIONS:
Procedure: Ultrasound guided transversus abdominis plane block — Using an 18 G Tuohy needle (80 mm Smiths medical Portex®) and the layers of the abdominal wall will be identified guided by superficial high-frequency 45 mm linear array ultrasound probe (13 MHz) as described by McDonnell and colleagues.(1) Twenty millilitre of 0.25% bupivacaine will be injected slowly after careful aspiration to ensure no vascular injury has occurred. Successful injection will produce an echo-lucent space between the muscle layers (internal oblique and transversus abdominis). All TAP blocks will be performed by the same anesthetist.

SUMMARY:
TAP block provided increased postoperative analgesia and reduced analgesic requirements as part of a multimodal analgesic regimen.

The aim of the study is to compare the efficacy of single low dose of intravenous MgSO4 versus intravenous dexamethasone as adjuvants to ultrasound guided TAP block for prolongation of postcesaren analgesia

DETAILED DESCRIPTION:
Study Setting: Ain shams University maternity Hospitals, Cairo, Egypt. Study Period: 4 months from 1st December 2019 to 1st April 2020. Sampling Method: Random sample Sample Size: 60 patients Study Design A total of (60) full term pregnant women (completed 37 weeks) will be recruited for the study will undergo elective cesarean section. Written informed consent will be obtained from all patients before randomization. Randomization will be done with the help of a computer generated list of numbers. Patients will be divided randomly and equally into three groups (20) Patients each. The first group patients will be assigned to magnesium sulphate group (M), the second group of patients will be assigned to dexamethasone group (D) and the third group will be assigned to placebo group (C). Group assignment, preparation and administration of drugs will be performed by a junior anesthetist who is neither involved nor interested by any means in the study. Blind grouping will be kept to all including the patients themselves, until the completion of study.

Preoperative Anesthetic Assessment All patients will be subjected to a thorough medical history, physical examination with thorough airway assessment, laboratory investigations (fasting blood sugar, kidney, liver function tests, serum electrolytes, coagulation profile, and electrocardiogram) preoperatively. They will be also counseled about the anesthetic management and potential complications of both surgery and anesthesia, and the explanations of numerical pain analogue scale (NAS) from 0-10. All these data will be documented.

Anesthetic Protocol All participants will be admitted to operating theatre (OR) induction area where patient identification is confirmed and an 18-gauge intravenous cannula will be inserted to all Participants. Participants in group (M) will receive 50 mg/kg MgSO4 in 100 ml isotonic saline intravenous (I.V) over 20 minutes prior to induction of general anesthesia by 30 minutes, participants in group (D) will receive 2 mg Dexamethasone in 100 ml isotonic saline IV while participants in group (C) will receive 100 ml isotonic saline IV (placebo) by the same route and over the same duration as control.

General anesthesia will be induced with intravenous propofol 2.0 mg/kg, succinyl choline 1.0 mg/Kg then they will be intubated orally which is fixed after confirmation of its place by capnography and auscultation. Anesthesia will be maintained by 2% sevoflurane in 100% oxygen then atracurium 0.1 mg/kg will be given for maintenance of muscle relaxation. After delivery of the fetus and placenta, 2 mg midazolam, 1 µg/kg fentanyl and 10 IU oxytocin (in 500 ml ringer solution) will be administrated. Immediately after completion of surgery, each patient will receive ultrasound guided bilateral ultrasound guided TAP blocks. After that muscle relaxant will be antagonized by 40 µg/kg neostigmine and 20 µg/kg atropine, then awake extubation will be done and the patients will be transferred to the recovery unit. All patients will be monitored all through the surgery by standard monitors including, electrocardiogram, the pulse oximeter, non-invasive blood pressure, and capnography.

TAP Block Technique Using an 18 G Tuohy needle (80 mm Smiths medical Portex®) and the layers of the abdominal wall will be identified guided by superficial high-frequency 45 mm linear array ultrasound probe (13 MHz) as described by McDonnell and colleagues.(1) Twenty millilitre of 0.25% bupivacaine will be injected slowly after careful aspiration to ensure no vascular injury has occurred. Successful injection will produce an echo-lucent space between the muscle layers (internal oblique and transversus abdominis). All TAP blocks will be performed by the same anesthetist.

Postoperative Analgesic Regimen It will start immediately on arrival to the recovery unit where all patients will receive 1 gm of Acetaminophen IV. After that all patients will continue on acetaminophen 1 gm/6 h IV and 5 mg Nalbuphine IV will be given if breakthrough pain develops during the first day postoperative.

Patients Assessment Patients will be transferred to Post-anesthesia care unit PACU and upon arrival to PACU, a pulse oximeter and Non-invasive blood pressure (NIBP) monitors will be attached to the patients. Discharge criteria from PACU will be stable vital signs, pain score less than or equal to 2, no nausea or vomiting, calm and alert patient.

ELIGIBILITY:
Inclusion Criteria:

* singleton full term pregnancy ( completed 37 weeks)
* undergoing elective cesarean section
* ASA I, II

Exclusion Criteria:

* patients with ASA physical status class III-IV,
* morbid obesity with BMI > 35 kg.m-2 at initial hospital visit
* neuro-axial anaesthesia
* severe pre-eclampsia,
* diabetes mellitus,
* cardiovascular disease,
* renal disease,
* hypermagnesemia,
* history of analgesic administration or intake during past 24 hours,
* chronic use of steroids therapy,
* urgent cesarean sections,
* multiple gestations,
* history of relevant drug allergy,
* any possibility of anticipated difficult intubation.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of postoperative analgesia | the first 24 hours postoperative
  pain assessed by visual analogue scale from 0- 10 as 0 means no pain and 10 worst pain and 0-3 mild pain , 4-7 moderate pain and 7-10 severe pain
The duration of analgesia before needing rescue analgesia | First 24 hours postoperative
  Time in minutes
Frequency of rescue analgesia needed | First 24 hours postoperative

SECONDARY OUTCOMES:
fetal safety | first minute and at 5 minutes postdelivery
  assessed by APGAR score from 1- 10 the higher the score the better the baby health a score of 7 to 9 means normal newborn and is a sign of good health after birth
time needed to ambulate unaided | the first 24 hours postoperatively
  Measured in hours
patient hemodynamics | Immediatelypre-anesthesia, immediately postintubation, immediately postextubation and 3o minutes postrecovery
  heart rate (BPM)
Patient hemodynamics | Immediatelypre-anesthesia, immediately postintubation, immediately postextubation and 3o minutes postrecovery
  Mean arterial blood pressure(mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams University, Faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No